CLINICAL TRIAL: NCT05848128
Title: A Phase 3, Multicenter, Randomized, Double-Masked, Vehicle-Controlled Clinical Study to Assess the Efficacy and Safety of 5% Tavilermide Ophthalmic Solution for the Treatment of Dry Eye
Brief Title: Efficacy and Safety Evaluation of Tavilermide Ophthalmic Solution for the Treatment of Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mimetogen Pharmaceuticals USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIM-729
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Dry Eye Syndromes; Dry Eye Disease; Kerato Conjunctivitis Sicca
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 5% Tavilermide ophthalmic solution (Experimental)
  Interventions: Drug: 5% Tavilermide ophthalmic solution
- Vehicle ophthalmic solution (Placebo Comparator)
  Interventions: Other: Vehicle ophthalmic solution

INTERVENTIONS:
Drug: 5% Tavilermide ophthalmic solution — Twice a day topicial dosing
  Arms: 5% Tavilermide ophthalmic solution
Other: Vehicle ophthalmic solution — Twice a day topical dosing
  Arms: Vehicle ophthalmic solution

SUMMARY:
The purpose of the study is to compare the efficacy and safety of 5% tavilermide ophthalmic solution to placebo for the treatment of the signs and symptoms of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject-reported history of dry eye disease in both eyes for at least 6 months;
* History of use of artificial tear eye drops for dry eye symptoms;
* Total score of ≥40 on SANDE;
* TFBUT;
* Corneal fluorescein staining;
* Lissamine green conjunctival staining;
* Schirmer's test score.

Exclusion Criteria:

* Have participated in a previous tavilermide (MIM-D3) study;
* Have clinically significant slit lamp findings at Visit 1;
* Have a history of lacrimal duct obstruction within 12 months of Visit 1;
* Have an uncontrolled systemic disease;
* Be a woman who is pregnant, nursing or planning a pregnancy;
* Be a woman of childbearing potential who is not using an acceptable means of birth control;
* Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 45 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-05-11 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Total Corneal Fluorescein Staining as Measured by the NEI Scale | Baseline to Day 85
  The National Eye Institute (NEI) scale is a standardized grading system of 0-3 was used for each of the 5 areas on each cornea (central, superior, temporal, nasal, and inferior). Grade 0 was specified when no staining is present. The maximum score was 15.
Change From Baseline in Eye Dryness Score as Measured by the VAS | Baseline to Day 85
  The Visual Analog Scale (VAS) where subjects were asked to rate their eye dryness (OU) by placing a vertical mark on the horizontal line to indicate their current level of discomfort. 0 mm corresponds to "No Discomfort," and 100 mm corresponds to "Maximal Discomfort." The length of the assessment line is 100 mm.

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Eye Doctors of Arizona, Phoenix, Arizona
  - Global Research Management, Glendale, California
  - LoBue Laser and Eye Medical Center, Murrieta, California
  - Eye Research Foundation, Newport Beach, California
  - Nature Coast Clinical Research, Crystal River, Florida
  - Eye Associates of Fort Myers, Fort Myers, Florida
  - Bowden Eye & Associates, Jacksonville, Florida
  - Shettle Eye Research, Largo, Florida
  - Eye Consultants of Atlanta, Atlanta, Georgia
  - Price Vision Group, Indianapolis, Indiana
  - Kannarr Eye Care, Pittsburg, Kansas
  - Seidenberg Protzko Eye Associates, Havre de Grace, Maryland
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - Silverstein Eye Centers, Kansas City, Missouri
  - Moyes Eye Center, Kansas City, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Rochester Ophthalmological Group, Rochester, New York
  - Oculus Research, Garner, North Carolina
  - James D. Branch, Winston-Salem, North Carolina
  - Abrams Eye Center, Cleveland, Ohio
  - Scott & Christie and Associates, Cranberry Township, Pennsylvania
  - West Bay Eye Associates, Warwick, Rhode Island
  - Total Eye Care, Memphis, Tennessee
  - Toyos Clinic, Nashville, Tennessee
  - Advanced Laser Vision & Surgical Institute, Houston, Texas
  - Lake Travis Eye & Laser Center/Revolution Research, Lakeway, Texas
  - PNV Clinical Research, San Antonio, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No